CLINICAL TRIAL: NCT04137705
Title: MultiOrgan Multi-Parametric MRI Study
Acronym: MORIS
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: CA0080
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multiparametric MRI — A standardised MRI protocol that provides a number of quantitative metrics on liver and other organs relevant to type 2 Diabetes - pancreas, kidneys, spleen, heart, lungs and aorta

SUMMARY:
To determine the reproducibility of a single quantitative multiparametric MRI for the assessment of body composition and multiple organ structures.

ELIGIBILITY:
Inclusion Criteria:

* Any person over 18 years of age.
* Participant is willing and able to give informed consent for participation in the investigation.
* EITHER: Participant has Type 2 Diabetes OR: Person is a healthy volunteer

Exclusion Criteria:

* The participant may not enter the investigation if they have any contraindication to magnetic resonance imaging (incl. pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the investigation, or may influence the result of the investigation, or the participant's ability to participate in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers, including healthy volunteers and individuals with Type 2 Diabetes (T2D).
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Assessment of repeatability (precision under the same conditions in the same subjects: 2 separate MRI acquisitions on the same scanner) of body composition and multiple organ metrics. | 24 months
  To determine the repeatability of multiparametric MRI in the assessment of body composition and multiple organ structures obtained within a single MR scanning session (liver, pancreas, aorta, heart, kidney, lungs and spleen)

SECONDARY OUTCOMES:
Assessment of the reproducibility (precision under different measurement conditions: same participants scanned on separate MRI scanners at both 1.5T and 3T) of multiparametric MRI for the assessment of body composition and multiple organ metrics. | 24 months
  To determine the reproducibility of multiparametric MRI in the assessment of body composition and multiple organ structures (liver, pancreas, aorta, heart, kidney, lungs and spleen) obtained within separate MR scanning sessions.

OTHER OUTCOMES:
Assessment of the mean differences in body composition and multiple organ metrics between healthy participants and those with type 2 diabetes acquired with multiparametric MRI. | 24 months
  To determine the range of body composition and multi-organ metrics (liver, pancreas, aorta, heart, kidney, lungs and spleen) in healthy participants and in those with type 2 diabetes assessed using multiparametric MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, Study Chair — Perspectum
Locations (3):
- United Kingdom (3):
  - Beaver House, Oxford
  - Oxford Centre for Magnetic Resonance, Oxford
  - Gemini One, Oxford